CLINICAL TRIAL: NCT04898452
Title: Intravenous Antibiotic Treatment at Home: A New Model for Across Services Interaction With the Use of Welfare Technology and Telemedicine.
Brief Title: Intravenous Antibiotic Treatment at Home
Acronym: Hosp@Home
Status: Recruiting | Type: Observational
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: SINTEF Health Research (Other); Kristiansund municipality (Unknown); Centre for Health Innovation (Unknown); Hospital Pharmacy of Central Norway Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019/60
Record Dates: First submitted 2020-07-01; First posted 2021-05-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Infection
Keywords: Home Care Services, Hospital-Based; Telemedicine; Home Infusion Therapy; Hospital at home; Antibiotics
MeSH Terms: conditions — Infections | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients needing antibiotics infusion: Patients needing antibiotics infusion A new model of interaction across health services with use of welfare technology and telemedicine Instead of admitted to the hospital, patients are followed up at home by the municipal regional response center and nurses in the response team according to the individual treatment plan. Hospital physicians are medically responsible throughout the course.
  Interventions: Other: A new model of interaction across health services with use of welfare technology and telemedicine
- Next of kin: Next of kin A new model of interaction across health services with use of welfare technology and telemedicine Instead of admitted to the hospital, patients are followed up at home by the municipal regional response center and nurses in the response team according to the individual treatment plan. Hospital physicians are medically responsible throughout the course.
  Interventions: Other: A new model of interaction across health services with use of welfare technology and telemedicine
- Health professionals: A new model of interaction across health services with use of welfare technology and telemedicine Instead of admitted to the hospital, patients are followed up at home by the municipal regional response center and nurses in the response team according to the individual treatment plan. Hospital physicians are medically responsible throughout the course.
  Interventions: Other: A new model of interaction across health services with use of welfare technology and telemedicine

INTERVENTIONS:
Other: A new model of interaction across health services with use of welfare technology and telemedicine — Instead of admitted to the hospital, patients are followed up at home by the municipal regional response center and nurses in the response team according to the individual treatment plan. Hospital physicians are medically responsible throughout the course.

SUMMARY:
The purpose of the study is to develop and evaluate a new model for across services interaction with the use of welfare technology and telemedicine. The model includes innovative and new routines for the exchange of patient information, quality systems and procedures between the municipality and the hospital. This model will first be tested for use in intravenous antibiotic therapy. The results of the study will be used to further develop the service. In the larger context, it is desirable to provide knowledge that is transferable to other diagnostic groups, treatment methods and geographical areas.

DETAILED DESCRIPTION:
This research-based innovation study has an evaluation approach with follow-up evaluation as the overall approach.

The pre-project was carried out with a qualitative approach under the auspices of SINTEF 2018/2019.

The main project consists of sub-study 1 and sub-study 2 (2020/2022).

Sub-study 1: The project use an iterative, user-centered service methodology with a qualitative approach. Here, SINTEF has the main responsibility for a qualitative summary after conducting interviews, observations and group discussions with patients, next of kins and health professionals regarding the development and testing / quality assurance of the new concept / service course for home treatment.

Sub-study 2: The approach here is quantitative. Descriptive data must be obtained from the hospital and municipal patient records, patient administration system (PAS) at Kristiansund hospital, alarm data from the Regional Response Center and pump log from the individual patient's infusion pump after home treatment.

ELIGIBILITY:
Inclusion criteria:

* Main or bi-diagnosis during stay:

A692 Borreliosis G00 - G009 Central nervous system inflammatory disorders I33 Endocarditis J86 Empyema D46.3 Spondylodiscitis M86 Osteomyelitis T84 Prosthesis / osteosynthesis infections M00.0-M00.9 Pyogen / septic arthritis J40-J47 Chronic diseases of the lower respiratory tract

* Competent to give consent
* The infection can not be treated with oral antibiotics in monotherapy
* Selected IV antibiotics must be suitable for administration via selected pumps
* The patient's condition is stable and does not require frequent observation by health care professionals
* The patient is motivated and willing to participate in intravenous treatment in home hospitals
* Must, after training, demonstrate mastery of practical procedures related to pump handling and any other procedures described in the patient's treatment plan
* The home must be suitable for intravenous antibiotic treatment; access to refrigerators, hygienic conditions, social conditions
* The patient must have a mobile phone and be able to handle the system for fast and secure communication with the Regional Response Center (RRO)

Exclusion criteria:

* consent not given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participate in both study part 1 (qualitative) and study part 2 (quantitative). Health professionals and next to kins participate in study part 1 (qualitative).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
number of rehospitalisations | 45 months
patient satisfaction | 45 months
  assessed with semi-structured interview
health personnel's opinion on patient safety | 45 months
  based on answers in web-case-registration-form (CRF)

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Hole, md phd, Study Director — Møre og Romsdal Hospital Trust
Locations (1):
- Helse Møre og Romsdal HF, Kristiansund sjukehus, Medisinsk Avdeling, Kristiansund, Norway